CLINICAL TRIAL: NCT06699459
Title: Irinotecan Liposomes +5-FU/LV or Capecitabine in Patients at High Risk of Recurrence After Resection of Resectable Biliary Tract Carcinoma: A Prospective Phase II Study
Brief Title: Irinotecan Liposomes +5-FU/LV Versus Capecitabine in Patients of Recurrence After Resection of Resectable BTC
Acronym: NICRRBTC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Zhejiang Cancer Hospital (Other); RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Fujian Provincial Hospital (Other); Ningbo No. 1 Hospital (Other); Shaoxing People's Hospital (Other); Southern Medical University, China (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH.20240559
Record Dates: First submitted 2024-11-13; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Biliary Tract Carcinoma
Keywords: Biliary Tract Carcinoma; Adjuvant treatment; Resectable; Irinotecan liposomes; Capecitabine
MeSH Terms: interventions — irinotecan sucrosofate; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan liposome (Experimental): * Irinotecan liposomes: 70mg/m2, intravenous infusion, Q2W, d1; ②LV: 400mg/m2, intravenous infusion, Q2W, d1; ③5-FU: 2400 mg/m2, continuous intravenous infusion, Q2W, d1-2;
  Interventions: Drug: Irinotecan Liposome
- Capecitabine (Other): Capecitabine, 1250mg/m2 oral, bid, Q3W, d1-14;
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Irinotecan Liposome — ②LV: 400mg/m2, intravenous infusion, Q2W, d1; ③5-FU: 2400 mg/m2, continuous intravenous infusion, Q2W, d1-2;
  Other Names: Irinotecan Liposome+LV/5-FU
  Arms: Irinotecan liposome
Drug: Capecitabine — ① Capecitabine, 1250mg/m2 orally, bid, Q3W, d1-14;
  Arms: Capecitabine

SUMMARY:
Irinotecan liposome combined with 5-FU/LV has shown good efficacy and has certain advantages in reducing the adverse reactions of conventional chemotherapy drugs. Adjuvant treatment of high-risk factors after surgery for biliary tract tumors can be further explored and attempted. Therefore, this study intends to conduct an exploratory study comparing oral capecitabine with irinotecan liposome +5-FU/LV for adjuvant therapy in high-risk patients after resection of resectable biliary malignancies, and evaluate the effectiveness and safety of irinotecan liposome +5-FU/LV as adjuvant therapy for high-risk patients after resection of resectable biliary malignancies. So it can provide more treatment options for patients with postoperative adjuvant therapy of biliary tract malignant tumor.

The DFS rate one year after surgery for biliary malignancy was assumed to be 51.4% with a maximum response rate of poor efficacy and 71.4% with a minimum response rate of good efficacy. A two-stage design was adopted with α=0.05 and certainty (1-β) =0.8, and Minimax was adopted. If a response occurs in 7 out of 14 patients or less, treatment options are rejected; In the second phase, if 24 or fewer responses occur in 38 patients, the protocol is rejected. A total of 38 samples were designed in two stages. The 1-year DFS rate was at least 65.8% in the total population of the test and control groups.

DETAILED DESCRIPTION:
According to the 2023 CSCO guidelines, differentiated surgical treatment has been performed for the site of biliary malignancies. For postoperative adjuvant therapy, BILCAP study showed that oral capecitabine as a single drug is one of the options for both efficacy and safety. For patients with postoperative risk factors, serum carcinoembryonic antigen (CEA) and CA19-9 are of some significance for monitoring recurrence, and often serve as precursors for clinical judgment of recurrence or progression. For people with high risk factors for recurrence and progression, adjuvant therapy intensity needs to be strengthened. Oral capecitabine can no longer meet the needs of this population, so patients need to be given intravenous chemotherapy in advance to control progression, recurrence or metastasis. In this case, metastatic first-line therapy is often used for early intervention. The NIFE study showed that compared with conventional chemotherapy regimens, the regimen of irinotecan liposome (new formulation) combined with 5-FU/LV achieved relatively better efficacy data in the median OS and ORR efficacy. It is noteworthy that this regimen has a significant therapeutic benefit in patients with advanced first-line extrahepatic cholangiocarcinoma, with a median PFS of 9.59 months and a median OS of 18.23 months.

To explore the efficacy and safety of irinotecan liposomes +5-FU/LV versus oral capecitabine in patients at high risk of recurrence after resection of resectable biliary malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old.
* Patients with histologically confirmed, resectable biliary malignancies with R0 resection.
* Postoperative pathology indicated the following risk factors: positive lymph nodes, vascular invasion, nerve invasion and so on.
* Has not received systemic chemotherapy before.
* The ECOG score is 0 to 1.
* Bone marrow and organ function were good: ① Neutrophils (ANC) ≥1.5×109/L, platelets (PLT) ≥100×109/L, hemoglobin (Hb) ≥90g/L, white blood cells (WBC) ≥3.0×109/L, albumin (ALB) ≥32 g/L, and no bleeding tendency; ② Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤2.5× upper limit of normal range (ULN), ≤5×ULN with liver metastasis; Total bilirubin ≤1.5×ULN; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 mL/min (calculated according to Cockroft-Gault).
* Expected survival ≥3 months.
* Volunteer to participate in the study and sign the informed consent. If the subject does not have the ability to read the informed consent (e.g., illiterate subjects), a witness must witness the informed process and sign the informed consent.

Exclusion Criteria:

* Patients allergic to the investigational drug and its excipients.
* Known or suspected central nervous system or lymphatic metastasis.
* Cannot discontinue use or has not discontinued use of CYP3A, CYP2C8, and UGT1A1 potent depressants or inducers (e.g., anticonvulsants [phenytoin, phenobarbital, or carbamazepine] within 2 weeks prior to enrollment), rifampicin, rifambutin, St.John's Wort, Grapefruit juice, clarithromycin, Itraconazole, Lopinavir, Nefazodone, Nelfinavir, Ritonavir, Saquinavir, Terrapivir, voriconazole, Azanavir, Gefilozil, Indinavir, etc.).
* There are signs and symptoms of intestinal obstruction.
* Other malignancies within the past 5 years or currently, except for cured cervical carcinoma in situ, uterine carcinoma in situ, and non-melanoma skin cancers.
* Autoimmune disease or long-term steroid use.
* Patients who are pregnant or nursing women, and patients who refuse to receive contraception during their reproductive age.
* Patients deemed unsuitable for participation in this study.
* Vulnerable groups, including people with mental illness, cognitive impairment, critically ill patients, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-11-14 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
one year DFS rate | From date of randomization until the date of one year
  The percentage of patients free of disease when the disease-free survival is at the 1-year node

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from initiation of treatment to first recording of PD or death
Overall survival | From date of randomization until the date of death from any cause, assessed up to 24 months
  The time between the start of treatment and the first recorded death
Disease-free survival | From date of randomization until the date of first tumor recurred or metastasized or date of death from any cause, whichever came first, assessed up to 24 months
  From randomization to the time when the first tumor recurred or metastasized, or when the subject died for any reason
adverse events | Incidence and severity of adverse events in treatment regimens up to 24 months
  Incidence and severity of adverse events in treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: Mingyu Chen, Ph.D, Principal Investigator — Sir Run Run Shaw Hospital
Locations (6):
- China (6):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital , affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Decide whether to share research data after publication